CLINICAL TRIAL: NCT06423248
Title: The Effect of Therapeutic Doses of Culinary Spices in Metabolic Syndrome: a Randomized Controlled Trial.
Brief Title: Culinary Spices in Metabolic Syndrome.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: United Arab Emirates University (Other)
Responsible Party: Principal Investigator, Ayesha Salem Al Dhaheri, Professor, Associate Provost, Student Affairs, United Arab Emirates University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Protocol Number: 15/22
Record Dates: First submitted 2024-05-15; First posted 2024-05-21 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2024-05

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome | interventions — ginger extract; Nigella sativa oil

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Both patient and investigators were blind to treatment allocation, with an independent researcher providing the allocated treatments to the participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Ginger (Active Comparator): 3g of dried powdered Ginger (Zingiber officinale) daily for 12 weeks.
  Interventions: Dietary Supplement: Ginger
- Cinnamon (Active Comparator): 3g of dried powdered Cinnamon (Cinnamomum) daily for 12 weeks.
  Interventions: Dietary Supplement: cinnamon
- Black Seed (Active Comparator): 3g of dried powdered Black Seed (Nigella sativa) daily for 12 weeks.
  Interventions: Dietary Supplement: black seed
- Placebo (Placebo Comparator): 3g of powdered corn starch daily for 12 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Ginger — 3g of dried powdered Ginger daily for 12 weeks
  Arms: Ginger
Dietary Supplement: black seed — 3g of dried powdered Black Seed daily for 12 weeks
  Arms: Black Seed
Dietary Supplement: cinnamon — 3g of dried powdered Cinnamon daily for 12 weeks.
  Arms: Cinnamon
Other: Placebo — 3g of powdered corn starch daily for 12 weeks.
  Arms: Placebo

SUMMARY:
This double blind, placebo controlled randomized controlled trial aims to evaluate the effect of three commonly used culinary spices - ginger (Zingiber officinale), cinnamon (Cinnamomum) and black seed (Nigella sativa) on the cardiometabolic parameters of individuals with risk factors of metabolic syndrome. Participants consume their assigned treatment for 12 weeks, and key cardiovascular and glucometabolic parameters are recorded at baseline, week 6, and week 12 of the study.

ELIGIBILITY:
Inclusion Criteria:

* age (18-50 years)
* 2 or more of MetS diagnostic criteria:
* high waist circumference (>80 cm for female and >94 cm for males),
* elevated blood pressure (equal to or greater than 130/85 mm Hg or use of medication for hypertension),
* high fasting blood glucose (equal to or greater than 100 mg/dL [5.6 mmol/L] or use of medication for hyperglycemia),
* lowered HDL cholesterol (less than 40 mg/dL [1.03 mmol/L] for men and less than 50 mg/dL [1.29 mmol/L] for women) and
* increased triglycerides (equal to or greater than 150 mg/dL [1.7 mmol/L]). Participants who had at least three risk factors out of five or had two risk factors and one borderline were included in the study.

Exclusion Criteria

* older than 50 years old or younger than 17 years old and
* did not meet the metabolic syndrome diagnostic criteria
* allergic to spices
* current smokers
* pregnant women
* lactating women or
* currently taking medication and if they
* refused to provide blood sample.
* acute illnesses
* chronic diseases such as kidney, liver, cardiovascular and gastrointestinal diseases were excluded from the study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2015-05-10 (Actual); Primary Completion 2016-11-13 (Actual); Study Completion 2016-11-13 (Actual)

PRIMARY OUTCOMES:
Mean Change in Fasting Blood Glucose at 12 weeks | Baseline, Week 6 and Week 12
  Fasting plasma glucose blood test taken at baseline, week 6 and week 12.
Mean Change in HbA1c at 12 weeks | Baseline, Week 6 and Week 12
  Glycated Haemoglobin blood test taken at baseline, week 6 and week 12.

SECONDARY OUTCOMES:
Mean Change in Blood Pressure at 12 weeks | Baseline, Week 6 and Week 12
  Systolic and diastolic blood pressure taken at baseline, week 6 and week 12.
Mean Change in Total Cholesterol at 12 weeks | Baseline, Week 6 and Week 12
  Total Cholesterol Blood Test taken at baseline, week 6 and week 12.
Mean Change in LDL Cholesterol at 12 weeks | Baseline, Week 6 and Week 12
  Low Density Lipoprotein Blood Test taken at baseline, week 6 and week 12.
Mean Change in HDL Cholesterol at 12 weeks | Baseline, Week 6 and Week 12
  High Density Lipoprotein Blood Test taken at baseline, week 6 and week 12.
Mean Change in Triglyceride concentrations at 12 weeks | Baseline, Week 6 and Week 12
  Triglyceride Blood Test taken at baseline, week 6 and week 12.
Mean Change in Weight at 12 weeks | Baseline, Week 6 and Week 12
  Weight taken at baseline, week 6 and week 12.
Mean Change in Body Mass Index at 12 weeks | Baseline, Week 6 and Week 12
  Weight taken at baseline, week 6 and week 12, and BMI calculated as weight divided by height squared.
Mean Change in Waist Circumference at 12 weeks | Baseline, Week 6 and Week 12
  Waist Circumference taken at baseline, week 6 and week 12.
Mean Change in Waist to Hip ratio at 12 weeks | Baseline, Week 6 and Week 12
  Waist and Hip Circumference taken at baseline, week 6 and week 12, and Waist-Hip ratio calculated.
Mean Change in Densitometric Body Composition at 12 weeks | Baseline, Week 6 and Week 12
  Dual Energy Xray Absorptiometry performed at baseline, week 6 and week 12, and Fat mass, body fat percentage, visceral fat, fat free mass, and skeletal muscle mass calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- United Arab Emirates University, Al Ain City, Abu Dhabi Emirate, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No